CLINICAL TRIAL: NCT07045467
Title: Pharmacokinetics and Pharmacodynamics of Continuous Infusion of Remimazolam in Kidney Transplant Recipients: A Multicenter Interventional Study
Brief Title: Remimazolam Infusion in Kidney Transplant Patients: A Multicenter Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Guanghan Wu, Department of Anesthesiology and Perioperative Medicine, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2024(103)
Record Dates: First submitted 2025-06-05; First posted 2025-07-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases; Renal Transplantation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All enrolled participants receive Remimazolam Besylate via continuous IV infusion (Experimental): All enrolled participants receive a standardized Remimazolam Besylate-based anesthesia protocol for renal transplant surgery, as follows:
  1. Intervention Drug:
     ◦ Remimazolam Besylate (Trade name: Rymazol®), supplied as a lyophilized powder (25 mg/vial) reconstituted with sterile water.
  2. Dosing Regimen:
     * Induction: Continuous IV infusion at 6 mg/kg/h until loss of consciousness (defined as MOAA/S score ≤1).
     * Maintenance: Titrated IV infusion (0.5-2 mg/kg/h) to maintain target anesthesia depth (Narcotrend Index: 27-60) until end of surgery.
  3. Ancillary Medications (per protocol §7.2):
     * Analgesia: Sufentanil (0.4-0.5 μg/kg induction; 10 μg at peritoneum closure) + Remifentanil infusion intraoperatively.
     * Muscle Relaxant: Rocuronium (0.6 mg/kg induction; 0.15 mg/kg bolus PRN).
     * Immunosuppression: Methylprednisolone 750 mg + Furosemide 60 mg pre-reperfusion.
     * Prohibited Agents: Sevoflurane, propofol, midazolam, dexmedetomidine, or etomidate.
  4. Depth Monitoring:
     * Real-time Narcot
  Interventions: Drug: Remimazolam Besylate

INTERVENTIONS:
Drug: Remimazolam Besylate — This is the first clinical trial evaluating Remimazolam's pharmacokinetics (PK), pharmacodynamics (PD), and safety in renal transplant recipients-a population with unique physiological alterations due to end-stage renal disease and graft reperfusion. Key differentiators include:
  Population-Specific Dosing Protocol:
  Induction: 6 mg/kg/h until MOAA/S ≤1 (vs. 5-12 mg/kg/h in general surgery).
  Maintenance: Titrated (0.5-2 mg/kg/h) to Narcotrend Index 27-60 (lower than typical BIS 40-60 targets), accounting for altered drug metabolism post-transplant.
  Transplant-Specific Context:
  Administered alongside standard immunosuppressants (methylprednisolone 750 mg + furosemide 60 mg at reperfusion) but prohibits common sedatives (midazolam/propofol) to isolate Remimazolam's effects.
  PK/PD sampling accounts for graft function dynamics (e.g., blood draws during reperfusion and post-op days 1-6).
  Exploratory Genetic Analysis:
  First study linking VDR/

SUMMARY:
The goal of this clinical trial is to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of remimazolam (CNS 70754) in healthy adult participants. The main questions it aims to answer are:

What are the key pharmacokinetic parameters of remimazolam, including peak concentration (Cmax), time to peak concentration (Tmax), area under the curve (AUC), and elimination half-life (T1/2)? What is the effect of remimazolam on consciousness, as measured by the MOAA/S scale and Narcotrend monitoring during anesthesia? Researchers will compare the pharmacokinetic and pharmacodynamic effects of remimazolam to see if the drug provides consistent and predictable sedation without significant adverse effects.

Participants will:

Receive continuous Infusion of Remimazolam. Have blood samples taken at various time points to measure plasma concentrations and calculate PK parameters.

Be monitored for consciousness and sedation levels using the MOAA/S scale and Narcotrend.

Undergo safety assessments, including laboratory tests, vital signs monitoring, and physical examinations throughout the study.

This study will help determine the drug's behavior in the body and its impact on sedation, providing valuable information for its future clinical use in anesthesia and other medical applications.

Last updated on December 22, 2024

ELIGIBILITY:
Inclusion Criteria Signed informed consent

Age ≥18 years and <65 years

Chronic renal failure scheduled for renal transplantation

Body mass index (BMI) 18-30 kg/m² (inclusive)

Weight ≥50 kg (males) or ≥45 kg (females)

ASA physical status classification III or IV

Exclusion Criteria Hepatic, psychiatric, or neurological disorders

Coagulopathy

Heart failure

Respiratory failure

Long-term sedative or antidepressant use

Pregnancy or lactation

Inability to communicate or cooperate

Participation in other drug/device trials within 3 months prior

Positive hepatitis B surface antigen (HBsAg)

Positive hepatitis C antibody (HCV-Ab)

Positive HIV antibody

Positive syphilis antibody

Use of hepatic enzyme inhibitors/inducers within 30 days prior (per Appendix 1)

Known hypersensitivity to ≥2 substances

Alcohol consumption >14 units/week within 6 months prior*

Drug abuse history within 3 months prior

Major infection/trauma within 1 month prior

Gastrointestinal surgery affecting drug absorption within 1 month prior

Vaccination within 1 month prior or planned during study

Blood loss/donation >400 mL within 3 months prior

Blood transfusion within 1 month prior

INR >1.5, PT >ULN+4 seconds, or APTT >15×ULN

Significant bleeding history within 3 months prior

Current anticoagulant therapy

Any condition deemed unsuitable by investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Remimazolam Plasma Concentration | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Blood concentration (ng/mL) of Remimazolam
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Maximum Plasma Concentration
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Area Under the Curve (0 to last measurable t)
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Area Under the Curve (0 to infinity)
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Time to Cmax
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Terminal Elimination Half-Life
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Total Body Clearance
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Renal Clearance
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Apparent Volume of Distribution (Terminal)
Remimazolam PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Mean Residence Time
Remimazolam PK Parameters | Pre-infusion, 2/5/10/20/30/45/60/120 minutes , hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes
  Percentage of AUC Extrapolated
CNS 7054 (Metabolite) PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Maximum Plasma Concentration
CNS 7054 (Metabolite) PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Area Under the Curve (0 to last measurable t)
CNS 7054 (Metabolite) PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Area Under the Curve (0 to infinity)
CNS 7054 (Metabolite) PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Time to Cmax
CNS 7054 (Metabolite) PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Terminal Elimination Half-Life
CNS 7054 (Metabolite) PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Mean Residence Time
CNS 7054 (Metabolite) PK Parameters | During surgery: Pre-infusion, 2/5/10/20/30/45/60/120 minutes, hourly until infusion stop; Post-infusion: 0/5/15/30/60/90/120/240 minutes.
  Percentage of AUC Extrapolated
Sedation Depth (PD) | Induction: every 1minutes until MOAA/S≤1; Maintenance: every 10 minutes; Recovery: every 2 minutes until 3 consecutive MOAA/S=5.
  MOAA/S score (0 to 5) + Narcotrend Index (NCI 0 to 100)
Time to Loss of Consciousness (MOAA/S ≤1) | 0 to 10 minutes after infusion start
  Time from infusion start to first MOAA/S score ≤1
Time to Full Alertness (3 consecutive MOAA/S=5) | Time from infusion stop to sustained alertness
  Time from infusion stop to sustained alertness
Narcotrend Index (NCI) Values | Continuous monitoring during infusion + 30 min post-stop
  Anesthesia depth index (0-100 scale)

SECONDARY OUTCOMES:
Postoperative Urine Output | Postoperation Days 1 to 6
  24-hour urine volume
Serum Creatinine Level | Preoperation, Postoperation Days 1 to 6
  Blood creatinine concentration
Estimated Glomerular Filtration Rate | Preoperation, Postoperation Days 1 to 6
  Kidney filtration rate
Intraoperative Hypotension Incidence | Intra-operative period
  MAP <65 mmHg for >1 minute
Intraoperative Bradycardia Incidence | Intra-operative period
  HR <45 bpm for >1 min
Injection Pain Incidence | During induction (0 to 10 minutes)
  Participant-reported pain during drug administration
Postoperative Nausea/Vomiting Incidence | PACU admission to Postoperation Day 6
  Postoperative Nausea/Vomiting occurrence
Postoperative Agitation Incidence | PACU stay (0 to 2 hours)
  RASS score ≥2
Delayed Recovery Incidence | End of surgery to PACU discharge
  Extubation time >30 min post-surgery
Intraoperative Awareness Incidence | Upon PACU discharge (Day 1)
  Positive Brice questionnaire response

OTHER OUTCOMES:
VDR Genotype Effect on Remimazolam Maximum Plasma Concentration | Pre-dose (Day 1)
  Correlation of VDR polymorphisms with peak concentration
CYP3A Genotype Effect on Remimazolam Area Under the Curve (0 to last measurable t) | Pre-dose (Day 1)
  Correlation of CYP3A polymorphisms with total exposure
POR Genotype Effect on Remimazolam Clearance | Pre-dose (Day 1)
  Correlation of POR polymorphisms with systemic clearance
VDR Genotype Effect on CNS 7054 Terminal Elimination Half-Life | Pre-dose (Day 1)
  Correlation of VDR polymorphisms with metabolite half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong First Medical University Hospital, Jinan, Shangdong, China